CLINICAL TRIAL: NCT01273779
Title: OASIS: A Phase 2/3 Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of Talactoferrin Alfa in Patients With Severe Sepsis
Brief Title: Safety and Efficacy of Talactoferrin Alfa in Patients With Severe Sepsis
Acronym: OASIS
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Data Safety Monitoring Board recommendation
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LF-0802
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Severe Sepsis
Keywords: sepsis; talactoferrin; lactoferrin; recombinant human lactoferrin
MeSH Terms: conditions — Sepsis | interventions — talactoferrin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Talactoferrin alfa (Experimental)
  Interventions: Drug: Talactoferrin alfa

INTERVENTIONS:
Drug: Talactoferrin alfa — 15 mL of an oral solution of 100mg/mL (1.5 g) given 3 times a day for up to 28 days or until discharge from the intensive care unit
  Arms: Talactoferrin alfa
Drug: Placebo — 15 mL of oral solution of placebo given 3 times a day for up to 28 days or until discharge from the intensive care unit
  Arms: Placebo

SUMMARY:
Study will evaluate the safety and potential benefit of talactoferrin (recombinant human lactoferrin) as an addition to the standard care for severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Onset of severe sepsis within the previous 24 hours
* Must be receiving antibiotic therapy
* Informed consent form signed by patient or authorized representatives according to local rules or regulations
* Able to take liquid medication by mouth or feeding tube

Exclusion Criteria:

* Receipt of investigational medication within 4 weeks prior to participation in the study
* Pregnant or breast-feeding
* Severe congestive heart failure
* Known severe HIV infection
* Presence of severe burns
* Patients on high dose immunosuppressants
* Patients whose death is considered imminent
* Patients whose life expectancy for concurrent illness is less than 6 months
* Severe hypoxic encephalopathy or persistent vegetative state
* Severe liver disease
* Chronically bed bound
* Patient, legal representative or patient's primary physician not committed to providing full, aggressive life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
All Cause Mortality | 28 Days

SECONDARY OUTCOMES:
All Cause Mortality | 3 months
All Cause Mortality | 6 months
All Cause Mortality | 12 months
Assess Safety and Tolerability | 28 days

CONTACTS AND LOCATIONS:
Locations (100):
- United States (34):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Maricopa Medical Center, Maricopa, Arizona
  - St. Joseph Hospital, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Stanford University Hospital, Stanford, California
  - UCLA Medical Center, Sylmar, California
  - Denver Health Medical Center, Denver, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Bay Area Chest Physicians, Clearwater, Florida
  - Eastern Idaho Medical Consultants, Idaho Falls, Idaho
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - Peoria Pulmonary Associates, Peoria, Illinois
  - Methodist Research Institute, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. Johns Mercy Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Moses Cone Memorial Hospital, Greensboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Cancer Institute, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - Texas Tech Health Science Center, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - LDS Hospital, Murray, Utah
  - University of Wisconsin Medical School, Madison, Wisconsin
- Belgium (10):
  - Clinique Saint-Pierre, Ottignies, Ottignies
  - Hôpitaux IRIS Sud, Brussels
  - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Gent, Ghent
  - CHU de Liège, Liège
  - Centre Hospitalier de Dinant, Mons
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir
- Canada (9):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - SMBD - Jewish General Hospital, Montreal, Quebec
- Denmark (2):
  - Aalborg Sygehus, Aalborg
  - Odense universitetshospital, Odense
- France (12):
  - Hôpital Universitaire Dupuytren, Limoges, Limoges
  - Hôtel Dieu, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Départemental La Roche sur Yon, Luçon, Montaigu - Les Oudaries, La Roche-sur-Yon
  - Hôpital Albert Michallon / La Tronche, La Tronche
  - Centre Hospitalier de Montauban, Montauban
  - Hôpital de la Source, Orléans
  - Hôpital Cochin, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Miletrie, Poitiers
  - Centre Hospitalier Angouleme, Saint-Michel
  - Hôpital Bretonneau, Tours
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Helios Klinikum Erfurt, Erfurt
  - Klinikum der Johann-Wolfgang Goethe-Universität, Frankfurt am Main
  - Klinikum der Friedrich-Schiller-Universität Jena, Jena
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Klinikum Harlaching, München
- Israel (6):
  - Rambam Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Western Galilee Hospital - Nahariya, Nahariya
  - Rabin Medical Center, Petah Tikva
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - VU Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - UMC St. Radboud, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
- Spain (9):
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitari De Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital de Sabadell, Sabadell, Catalonia
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Catalonia
  - Hospital Mutua de Terrassa, Terrassa, Catalonia
  - Hospital Clinico San Carlos, Madrid, Madrid, Communidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Communidad de
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario La Paz, Madrid
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - St James's University Hospital, Leeds
  - St John's Hospital, Livingston
  - University College London, London
  - St. Thomas' Hospital, London

REFERENCES:
- [Derived] Vincent JL, Marshall JC, Dellinger RP, Simonson SG, Guntupalli K, Levy MM, Singer M, Malik R; Oral tAlactoferrin in Severe sepsIS Study Investigators. Talactoferrin in Severe Sepsis: Results From the Phase II/III Oral tAlactoferrin in Severe sepsIS Trial. Crit Care Med. 2015 Sep;43(9):1832-8. doi: 10.1097/CCM.0000000000001090. PMID 26010687